CLINICAL TRIAL: NCT00461552
Title: Therapeutic Approaches to HAART-Induced Lipodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Abhimanyu Garg, Chairman, Division Nutrition and Metabolic Diseases, Professor Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 063656
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: Lipodystrophy; HIV; HAART; HIV Lipodystrophy Syndrome; Lipodystrophy syndrome; HIV-Associated Lipodystrophy; HIV-Associated Lipodystrophy Syndrome; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy; HIV-Associated Lipodystrophy Syndrome | interventions — Leptin; metreleptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Leptin (Active Comparator): Leptin weight and gender based dose, sub-cutaneous, twice daily. Leptin versus placebo for entire 6 months double-blind.
  Interventions: Drug: Leptin
- Placebo (Placebo Comparator): Placebo , sub-Q injection twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Leptin — weight based, sub-cutaneous injection, twice daily
  Other Names: Metreleptin
  Arms: Leptin
Other: Placebo — weight based, sub-cutaneous injection, twice daily
  Arms: Placebo

SUMMARY:
To determine the efficacy and safety of 4 therapeutic interventions on HAART-Induced lipodystrophy. The interventions are: 1) Dietary - the effect of a high carbohydrate vs.a high cis-monounsaturated fatty acid diet. 2) The effect of aerobic exercise with dietary advice. 3) The effect of Omega-3 Fish Oil Capsules. 4) The effect of leptin therapy. These interventions are aimed at improving the metabolic complications of HAART therapy such as elevated lipids, and insulin resistance or diabetes.

DETAILED DESCRIPTION:
Patients with HAART-induced lipodystrophy report loss of subcutaneous (sc) fat from the extremities and face and excess fat accumulation in the neck and truncal region. They also are predisposed to metabolic complications of insulin resistance, such as, dyslipidemia and diabetes mellitus. The pathogenesis of HAART-induced lipodystrophy is not fully understood although PIs have been strongly implicated as the cause. The metabolic complications pose an increased risk of atherosclerosis and acute pancreatitis whereas changes in body fat distribution cause physical discomfort and psychological distress. Management of these problems poses a therapeutic challenge. We propose potentially safe therapeutic lifestyle changes as well as novel therapies for management of HAART-induced lipodystrophy and its metabolic complications. The hypotheses to be tested and the aims are:

Hypothesis 1: A diet rich in cis-monounsaturated fatty acids improves HAART-induced glucose intolerance and dyslipidemia in HIV-infected patients.

Aim 1: To compare acceptability and effects of isocaloric diets rich in carbohydrates and cis-monounsaturated fats, each given for 6 wk, on glucose and lipid metabolism in patients with HAART-induced dyslipidemia in a randomized, cross-over study.

Hypothesis 2: A regimen of aerobic exercise improves insulin resistance, dyslipidemia and body fat distribution in HIV-infected patients with HAART-induced lipodystrophy.

Aim 2: To determine the effects of a supervised aerobic exercise regimen and dietary advice on glucose and lipid metabolism, and body fat distribution in HIV-infected patients with HAART-induced lipodystrophy.

Hypothesis 3: The n-3 polyunsaturated fats improve HAART-induced dyslipidemia in HIV-infected patients.

Aim 3: To determine the lipid-lowering effects of n-3 polyunsaturated fats in a randomized, double-blind, placebo-controlled, crossover trial in HIV-infected patients with HAART-induced dyslipidemia.

Hypothesis 4: Leptin replacement improves insulin resistance, dyslipidemia and body fat distribution in patients with HAART-induced lipodystrophy and hypoleptinemia.

Aim 4 To study efficacy and safety of recombinant methionyl leptin (r-metHuleptin) in improving insulin sensitivity, dyslipidemia and body fat distribution in patients with HAART-induced lipodystrophy and hypoleptinemia using a randomized, double-blind, placebo-controlled, parallel design.

Results from these studies may help in designing therapeutic approaches to HAART-induced lipodystrophy and its metabolic complications as well as for prevention of these problems in HIV-infected patients being placed on HAART.

We are only reporting the results of Aim 4 - (Leptin Study) here.

ELIGIBILITY:
Inclusion Criteria - General inclusion:

* Age > 14 years
* HIV infection being treated with HIV-1 protease inhibitors for >6 months currently, or previous protease inhibitor therapy of at least 2 years duration with development of lipodystrophy and current stable therapy preferably for past 4 months.
* Fasting serum triglycerides > 200 mg/dL

Exclusion Criteria - General exclusion:

* Acute, ongoing AIDS-defining opportunistic infections.
* Blood CD4 positive lymphocyte count < 200/mm3
* Known liver disease due to causes other than nonalcoholic steatohepatitis with elevation of liver transaminases by more than two and a half times above the upper limits of normal (SGOT>105 U/L, SGPT>120 U/L) or total bilirubin (>1.5 mg/dL).
* Hematocrit of less than 30%.
* Current alcohol abuse (>7 drinks or 210 g per wk for women and >14 drinks or 420 g per wk for men).
* Current substance abuse.
* Uncontrolled diabetes mellitus with fasting plasma glucose > 180 mg/dL or hemoglobin A1c > 9%.
* History of weight loss during the last 3 months.
* Use of anorexiogenic drugs, thiazolidinediones, anabolic steroids and human growth hormone.
* Major Neuro-psychiatric illnesses impeding competence or compliance.
* Pregnant and lactating women.
* Cancer excluding skin cancer other than melanoma.
* Acute medical illnesses precluding participation in the studies.
* Chronic renal insufficiency with serum creatinine > 2 mg/dL.
* Untreated thyroid disorders such as hypothyroidism and hyperthyroidism. Each of the 4 treatment arms has additional specific inclusion and exclusion criteria

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, M.D., Principal Investigator — Univeristy of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Leptin: Randomized to receive leptin.
- Placebo: Randomized to receive placebo
Period: Overall Study
Arm/Group | Leptin | Placebo
Started | 7 | 7
Completed | 7 | 5
Not Completed | 0 | 2
Not completed — Drug Dispensing error | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leptin | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (10.4) | 48.1 (3.7) | 49.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Body Weight [Mean (Standard Deviation); unit: kg] | 71.2 (6.2) | 75.6 (7.8) | 73.4 (7.2)
Triglycerides [Median (Full Range); unit: mg/dL] | 336 [245 to 587] | 471 [238 to 1424] | 377 [238 to 1424]

OUTCOME MEASURES:

1. Primary Outcome: Fasting Serum Triglycerides
Time Frame: 6 months
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Leptin | Placebo
Number analyzed (Participants) | 7 | 5
mg/dL | 237 [122 to 439] | 341 [127 to 1099]
Statistical Analysis 1: Comparison: Leptin vs Placebo; Test type: Superiority; p = 0.84, Mixed Models Analysis — Treatment time month interaction

2. Secondary Outcome: Body Weight (kg)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Leptin | Placebo
Number analyzed (Participants) | 7 | 5
kg | 68.6 (5.7) | 73.3 (6.7)
Statistical Analysis 1: Comparison: Leptin vs Placebo; Test type: Other; p = 0.4, Mixed Models Analysis — Treatment time month interaction

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Leptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/5
Other Adverse Events (participants affected / at risk) | 4/7 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leptin (N=7) | Placebo (N=5)
cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) — Mild cerebrovascular event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leptin (N=7) | Placebo (N=5)
Itching (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) — Occasional itching, burning or bruising with injections

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days